CLINICAL TRIAL: NCT03098225
Title: A Phase IV, Randomized, Multi-center Clinical Trial to Compare the Efficacy of Orbital Radiotherapy in Association With Intravenous Glucocorticoids vs Intravenous Glucocorticoids Alone for Moderately Severe and Active Graves' Orbitopathy
Brief Title: A Trial to Evaluate the Efficacy of Orbital Radiotherapy in Graves' Orbitopathy
Acronym: ORGO
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pisa (Other)
Responsible Party: Principal Investigator, Marinò Michele, Ricercatore (Assistant Professor), University of Pisa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ORGO
Record Dates: First submitted 2017-03-21; First posted 2017-03-31 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Thyroid Associated Ophthalmopathy
MeSH Terms: conditions — Graves Ophthalmopathy | interventions — Methylprednisolone

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Ophthalmology blinded to treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Radiotherapy (Experimental): Patients with moderately severe GO treated with Intravenous glucocorticoids associated with orbital radiotherapy
  Interventions: Radiation: Orbital radiotherapy; Drug: Methylprednisolone
- No Radiotherapy (Active Comparator): Patients with moderately severe GO treated with Intravenous glucocorticoids alone
  Interventions: Drug: Methylprednisolone

INTERVENTIONS:
Radiation: Orbital radiotherapy — A high-voltage linear accelerator will be used and a cumulative radiation dose of 20 Gy will be delivered to each eye in 10 fractionated doses over a period of 2 weeks. All patients will be treated in both eyes.
  Other Names: OR
  Arms: Radiotherapy
Drug: Methylprednisolone — Methylprednisolone pulse therapy for 12 weeks as follows: 500 mg IV once weekly for 6 weeks, then 250 mg IV once weekly for a further 6 weeks. Cumulative dose 4.5 g.
  Other Names: ivGC

SUMMARY:
Graves' orbitopathy (GO) is a disfiguring and disabling disease that profoundly impairs the quality of life of affected patients. High dose intravenous (iv) glucocorticoids (GC) (ivGC) is a well established, widely used treatment for active GO. The use of systemic glucocorticoids takes advantage from their immune suppressive and antiinflammatory actions, resulting in an overall beneficial effect ranging from ~35 to ~60% of patients in various studies. The intravenous route of administration has been shown to be superior to the oral route, both in terms of GO outcome and side effect profile. The combination of ivGC and orbital radiotherapy (OR) is used routinely in patients with moderate-severe, active GO, as a second-line treatment, as also recommended in the recent Guidelines published by the European Thyroid Association/European Group on Graves' Orbitopathy. Thus, the majority of studies have shown that OR increases the response rate to GC. Those studies were performed using oral GC, whereas it is not known whether OR potentiate also the effects of ivGC.

The present study is aimed at determining whether OR potentiate the effects of ivGC in the treatment of moderately severe and active GO, in terms of GO outcome and quality of life. A possible extension of the study can be foreseen, aimed at investigating the very long time GO outcome.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of Graves' disease based on the presence of hyperthyroidism (either untreated or treated with antithyroid drugs) associated with detectable anti-TSH receptor autoantibodies
2. No major treatments for hyperthyroidism (thyroidectomy or radioiodine) in the last 3 months
3. Euthyroidism on anti-thyroid medications or L'thyroxine (LT4) since at least 2 months
4. GO symptoms lasting since no more than one year
5. Active GO: CAS ≥ 3 out of 7 (worst eye)
6. Moderate or moderately severe GO: at least one of the following signs (worst eye):

   * Exophthalmos ≥ 22 mm
   * Eye muscle involvement with mono-ocular ductions in any direction of gaze of less than 30° or evident dismotility
   * Diplopia according to Gorman score of grades a-c
7. No corticosteroids or immunosuppressive treatment for GO in the last 3 months
8. No contraindication to OR: diabetes, hypertension, retinopathy of any type, glaucoma
9. Male and female patients of age: 35-75 years
10. Effective method of contraception during the whole trial and at least six weeks after last intake of trial drugs (only female of reproducing age)
11. No mental illness that prevent patients from comprehensive, written informed consent
12. Compliant patient, regular follow-up possible

Exclusion Criteria:

1. Absence of Graves' hyperthyroidism (present or past)
2. Thyroidectomy or radioiodine in the last 3 months
3. Uncontrolled hyperthyroidism or hypothyroidism
4. GO symptoms lasting since more than one year
5. CAS <3 (worst eye)
6. Optic neuropathy
7. Contraindications to OR (diabetes, retinopathy of any kind)
8. Pregnancy, breast-feeding women
9. No informed consent
10. Acute or chronic liver disease
11. Relevant Malignancy
12. Chronic renal failure or other diseases of any relevance to prevent steroid treatment 13) Corticosteroids or other immunosuppressive agents within last 3 months
13. Recent (≤1 year) history of alcoholism or drug abuse
14. Previous orbital disease other than GO, eye injuries or surgery

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of overall GO outcome determined using a composite evaluation | 52 weeks
  A composite evaluation of GO was described previously.
  Improvement is defined as amelioration of two parameters in at least one eye, without deterioration of any parameters in both eyes:
  Deterioration is defined as worsening in two parameters in at least one eye:
  All other cases are defined as "no change"
  The parameters are:
  * Eyelid swelling (improvement/worsening according to EUGOGO Atlas evaluation)
  * Lid aperture in mm (significant variation: 2 or more mm)
  * Clinical activity score (CAS) (7 items: spontaneous pain, evoked pain, eyelid edema, eyelid redness, conjunctiva redness, caruncle edema, chemosis; significant change: at least 2 points)
  * Exophthalmos in mm (significant variation 2 or more mm)
  * Eye muscle involvement - diplopia score (Gorman score) (significant variation: disappearance or change in the degree, or improvement of ≥12 degrees in motility)

SECONDARY OUTCOMES:
Comparison of overall GO outcome determined using a composite evaluation | 26 weeks
  A composite evaluation of GO was described previously.
  Improvement is defined as amelioration of two parameters in at least one eye, without deterioration of any parameters in both eyes:
  Deterioration is defined as worsening in two parameters in at least one eye:
  All other cases are defined as "no change"
  The parameters are:
  * Eyelid swelling (improvement/worsening according to EUGOGO Atlas evaluation)
  * Lid aperture in mm (significant variation: 2 or more mm)
  * Clinical activity score (CAS) (7 items: spontaneous pain, evoked pain, eyelid edema, eyelid redness, conjunctiva redness, caruncle edema, chemosis; significant change: at least 2 points)
  * Exophthalmos in mm (significant variation 2 or more mm)
  * Eye muscle involvement - diplopia score (Gorman score) (significant variation: disappearance or change in the degree, or improvement of ≥12 degrees in motility)
Comparison of a disease specific quality of life questionnaire (GO-QoL) | 26 weeks
  Comparison of a disease specific quality of life questionnaire (GO-QoL)
GO relapse | 52 weeks
  GO worsening in comparison with the 26 week evaluation, by a composite GO score:
  Worsening is defined as worsening in two parameters in at least one eye:
  The parameters are:
  * Eyelid swelling (worsening according to EUGOGO Atlas evaluation)
  * Lid aperture in mm (significant worsening: 2 or more mm)
  * Clinical activity score (CAS) (7 items: spontaneous pain, evoked pain, eyelid edema, eyelid redness, conjunctiva redness, caruncle edema, chemosis; significant worsening: at least 2 points)
  * Exophthalmos in mm (significant worsening: 2 or more mm)
  * Eye muscle involvement - diplopia score (Gorman score) (significant worsening: appearance or change in the degree, or worsening of ≥12 degrees in motility)
Comparison of a disease specific quality of life questionnaire (GO-QoL) | 52 weeks
  Comparison of a disease specific quality of life questionnaire (GO-QoL)

IPD SHARING:
Plan to Share IPD: No